CLINICAL TRIAL: NCT05495048
Title: Transvaginal Natural Orifice Specimen Extraction Surgery Versus Conventional Laparoscopic Surgery With Mini-laparotomy in Right Hemicolectomy for Colon Cancer: a Randomised, Controlled, Phase 3, Non-inferiority Trial (NOSES VIIIA Trial)
Brief Title: Transvaginal NOSES Versus Conventional Laparoscopic Surgery for Right Hemicolectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Principal Investigator, Cai Zhenghao, Dr., Shanghai Minimally Invasive Surgery Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOSES VIIIA Trial
Record Dates: First submitted 2022-08-09; First posted 2022-08-10 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NOSES VIIIA (Experimental): totally laparoscopic right hemicolectomy with transvaginal natural orifice specimen extraction
  Interventions: Procedure: NOSES VIIIA
- laparoscopic surgery with mini-laparotomy (Active Comparator): laparoscopic right hemicolectomy with trans-abdominal extraction from a mini-laparotomy
  Interventions: Procedure: laparoscopic surgery with mini-laparotomy

INTERVENTIONS:
Procedure: NOSES VIIIA — totally laparoscopic right hemicolectomy with transvaginal natural orifice specimen extraction
  Arms: NOSES VIIIA
Procedure: laparoscopic surgery with mini-laparotomy — laparoscopic right hemicolectomy with trans-abdominal extraction from a mini-laparotomy
  Arms: laparoscopic surgery with mini-laparotomy

SUMMARY:
It is controversial that totally laparoscopic right hemicolectomy with transvaginal natural orifice specimen extraction (NOSES VIIIA) can provide non-inferior oncological outcomes compared to conventional laparoscopic surgery with mini-laparotomy in the treatment of right colon cancer. We aim to carry out a multicenter, open-lable, parallel, non-inferiority, phase III, randomized controlled clinical trial, which enrolls 356 female patients with cT1-3NxM0 right colon adenocarcinoma. They are randomly assigned to the experimental group (NOSES VIIIA) or the control group (laparoscopic surgery with mini-laparotomy) in a 1:1 ratio. Perioperative indicators, pathological results, quality of life and cosmetic evaluation will be compared between the two groups. Then, a three-year follow-up of these patients will provide evidence for long-term oncological outcomes of NOSES VIIIA.

ELIGIBILITY:
Inclusion Criteria:

* volunteer to participate and the informed consent signed;
* 18-75 years;
* female who have given birth;
* pathologically confirmed adenocarcinoma/high-grade intraepithelial neoplasia by preoperative colonoscopy and biopsy;
* preoperative CT or MRI indicates that the tumor diameter is no more than 5.0 cm;
* preoperative staging cT1-3NanyM0
* body mass index <30 kg/m2;
* willing to undergo laparoscopic right hemicolectomy

Exclusion Criteria:

* contraindications for laparoscopic surgery;
* emergency surgery due to acute intestinal obstruction, perforation or bleeding;
* distant metastasis;
* multiple colorectal cancer;
* has received preoperative chemoradiotherapy;
* with a history of other malignant tumors;
* unwilling to sign the informed consent or receive follow-up according to the study protocol.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
disease-free survival rate | 3 years after surgery
  disease-free survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, China

REFERENCES:
- [Derived] Yu M, Cai Z, Zhou H, Fingerhut A, He Z, Xue P, Song H, Yang X, Cheng X, Zhang S, Xu X, Zhong H, Abuduaini N, Liu J, Wang X, Feng B. Natural orifice specimen extraction surgery versus small-incision assisted laparoscopic radical right hemicolectomy. Future Oncol. 2023 Dec;19(40):2641-2650. doi: 10.2217/fon-2023-0769. Epub 2023 Dec 18. PMID 38108112